CLINICAL TRIAL: NCT05508022
Title: Determination of the Effect of Breathing Exercise Technique Applied to Children Aged 6-12 Before Enema on Anxiety, Fear and Pain
Brief Title: Determining the Effect of Breathing Exercise Applied to Children Aged 6-12 Before Enema on Anxiety, Fear and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Figen Türkdüdükçü, Doctor Lecturer, KTO Karatay University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KaratayUF
Record Dates: First submitted 2022-08-16; First posted 2022-08-19 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Constipation; Distention; Child, Only
Keywords: Children; Enema; Anxiety; Fear; Pain; Breathing exercise
MeSH Terms: conditions — Constipation; Dilatation, Pathologic; Anxiety Disorders; Pain | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: The research groups consisted of 106 (per group: 53) children who met the sample selection criteria. Children were randomly assigned to intervention and control groups. Assignment of children to groups was done by an independent statistician to ensure confidentiality and avoid bias. In this study, stratified randomization method was used to assign children to groups. In randomized controlled experimental studies, the number of cases in each group is required to be balanced and similar in terms of prognostic factors (such as age and gender). With the stratified randomization method, differences and undesirable situations between study groups are tried to be minimized. The permutation method is used to achieve this balance (Kahan ve ark., 2015). In this study, children were stratified according to age (6-9 and 10-12) and gender (female, male) variables.
Masking Description: Blinding of the participants and the nursing researcher who delivered the intervention was not possible due to the nature of the intervention. Veri toplama sürecinde yanlılığı önlemek için; lavman işleminden önce ve sonra klinkte çalışan bağımsız bir gözlemci hemşire tarafından ölçekler uygulandı. Before data collection, randomization was performed by the statistician by coding the intervention and control groups as "A" and "B". Analysis of the data was performed by a statistician to avoid bias in the evaluation of the data. After analyzing and interpreting the data during the statistical process, the codes of the intervention and control groups of the study were revealed. The statistician was blinded during the analysis of study data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breathing Exercise (Experimental): Breathing exercises will be applied to the participants in the experimental group.
  Interventions: Behavioral: Breathing exercise

INTERVENTIONS:
Behavioral: Breathing exercise — Before the enema is applied, breathing exercises will be applied to the participants in the intervention group.

SUMMARY:
In this study, it was aimed to determine the effect of breathing exercise applied before the enema procedure, which causes fear, pain and anxiety in children aged 6-12 years who applied to the pediatric emergency service, on fear, pain and anxiety in children. This research is in pretest-posttest, parallel group, randomized controlled experimental design.

The universe of the research consists of children aged 6-12 years who applied to the pediatric emergency department of Iğdır State Hospital (Turkey) between May 2022 and June 2022.

DETAILED DESCRIPTION:
In this study, it was aimed to determine the effect of breathing exercise applied before the enema procedure, which causes fear, pain and anxiety in children aged 6-12 years who applied to the pediatric emergency service, on fear, pain and anxiety in children. This research is in pretest-posttest, parallel group, randomized controlled experimental design.

The universe of the research consists of children aged 6-12 years who applied to the pediatric emergency department of Iğdır State Hospital (Turkey) between May 2022 and June 2022.

In the study, the pre-test scores of the pain, fear and anxiety levels of the children were compared and it was found that the pain, fear and anxiety levels of the intervention and control groups were moderate, and there was no difference between the groups. This result is important in terms of evaluating the effectiveness of the initiative.

In the study, a significant difference was found between the pain, fear and anxiety levels of the intervention and control groups after breathing exercise. Accordingly, the pain, fear and anxiety levels of the intervention group were significantly lower than the control group.

ELIGIBILITY:
Inclusion Criteria:

* Being between 6-12 years of age
* Administering an enema because of constipation or distension
* There should be no obstacle to the enema procedure
* Child and parent agree to participate in the study

Exclusion Criteria:

* Having a mental disability
* Having any problems with hearing, vision, hearing
* Taking analgesics within the last 6 hours
* Having an additional illness that may cause pain

Removal criteria were as follows:

* Developing complications during the enema procedure (intestinal perforation, bleeding, etc.)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Comparison of the anxiety level of the experimental group in which breathing exercise was applied | 20 minutes
  Before the enema application, the participants in the experimental group will be given breathing exercises. Thus, it is aimed to prevent the child from experiencing anxiety that may result from enema application. With this application, the effect of breathing exercise on anxiety will be monitored.
Comparison of the fear level of the experimental group in which breathing exercise was applied. | 20 minutes
  Before the enema application, the participants in the experimental group will be given breathing exercises. Thus, it is aimed to prevent the child from experiencing fear that may arise from enema application. With this application, the effect of breathing exercise on fear will be monitored.
Comparison of the pain level of the experimental group in which breathing exercise was applied | 20 minutes
  Before the enema application, the participants in the experimental group will be given breathing exercises. Thus, it is aimed to prevent the child from experiencing pain that may result from enema application. With this application, the effect of breathing exercise on pain will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Padir, Msc, Study Chair — Igdır State Hospital, Turkey
Locations (1):
- Kto Karatay University, Konya, Turkey (Türkiye)

REFERENCES:
- See also: Comparing the Effect of Two Methods of Distraction on the Pain Intensity Venipuncture in School-age Children: A Randomized Clinical Trial — https://ijp.mums.ac.ir/article_11038.html
- See also: Constipation and paediatric emergency department utilization — https://pubmed.ncbi.nlm.nih.gov/29479200/
- See also: Association between abdominal pain and fecal impaction grade assessed through radiography in constipated patients at a pediatric emergency service — https://pubmed.ncbi.nlm.nih.gov/31495541/
- See also: Soap Suds Enemas Are Efficacious and Safe for Treating Fecal Impaction in Children With Abdominal Pain — https://pubmed.ncbi.nlm.nih.gov/26655947/
- See also: Developing a New One-Dimensional Scale to Measure Pain in Children: Pencil Pain Scale — https://www.innovationinfo.org/journal-of-pediatrics-and-infants/article/Developing-a-New-One-Dimensional-Scale-to-Measure-Pain-in-Children-Pencil-Pain-Scale
- See also: The Effect of Breathing Exercise Using Bubble Blower on Anxiety and Pain during Inferior Alveolar Nerve Block in Children Aged 7 to 10 Years: A Crossover Randomized Clinical Trial — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8786543/
- See also: The effectiveness of a health promotion and stress-management intervention program in a sample of obese children and adolescents — https://pubmed.ncbi.nlm.nih.gov/30099726/
- See also: Effects of breathing exercise techniques on the pain and anxiety of burn patients: A systematic review and meta-analysis — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10333038/
- See also: Relaxation-guided imagery reduces perioperative anxiety and pain in children: a randomized study — https://pubmed.ncbi.nlm.nih.gov/30944985/
- See also: Effects of virtual reality on pain, fear and anxiety during blood draw in children aged 5-12 years old: A randomised controlled study — https://pubmed.ncbi.nlm.nih.gov/31889358/
- See also: The Effects of Cartoon Assisted Endoscopy Preparation Package on Children's Fear and Anxiety Levels and Parental Satisfaction in Turkey — https://pubmed.ncbi.nlm.nih.gov/32173165/
- See also: Soap bubbles as a distraction technique in the management of pain, anxiety, and fear in children at the paediatric emergency room: A pilot study. — https://europepmc.org/article/med/30466144
- See also: Medical management of constipation — https://pubmed.ncbi.nlm.nih.gov/23449608/
- See also: Psychosocial factors impacting antegrade continence enema outcomes in pediatric patients — https://pubmed.ncbi.nlm.nih.gov/37427680/